CLINICAL TRIAL: NCT06157346
Title: Characteristics of Intestinal Bacteria and Their Effects on Growth and Immune Function in Children at High Altitude in Diqing Tibetan Autonomous Prefecture, Yunnan Province
Brief Title: Characteristics of Intestinal Bacteria and Their Effects on Growth and Immune Function in Children at High Altitude
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SYJQ-001
Record Dates: First submitted 2023-11-08; First posted 2023-12-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Health; Children, Only; Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — faeces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-altitude: Children live in a high-altitude area of more than 3000 meters.
- Low-altitude: Children live in a low-altitude area of less than 500 meters.

SUMMARY:
Microbes and the human body maintain a complex relationship of interaction and influence. Different regions, altitudes, and dietary habits have different degrees of influence on the composition of children's intestinal flora. Therefore, the development and maturation process of children's intestinal flora in plateau areas was discovered, and its relationship with children's immunity, metabolism, and growth was understood. The mechanism of action of children's intestinal flora on immunity, growth and development was further analyzed by comparing it with people in low-altitude areas, to provide a scientific basis for improving children's health in plateau areas.

DETAILED DESCRIPTION:
This observational study aims to gain a deeper understanding of the interactions and influence of microbes on the human body. By comparing the gut microbiota composition of children in different regions, at varying altitudes, and with distinct dietary habits, the study aims to answer two key questions:

What are the characteristics of children's gut microbiota in different regions, at different altitudes, and with different dietary habits? What is the relationship between the development and maturation process of children's gut microbiota in plateau areas and their immunity, metabolism, and growth? Participants will be asked to provide fecal samples for analysis during the study. They may also be asked to answer questionnaires about their lifestyle factors such as diet and physical activity. The comparison group is included, researchers will compare the gut microbiota composition and diversity of children in low-altitude areas with those in plateau areas to assess any differences in their gut microbiota profiles. By comparing these differences, the mechanism of action of children's gut microbiota on immunity, growth and development can be further analyzed. The findings of this study aim to provide a scientific basis for improving children's health in plateau areas.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-3 years old
* Both men and women;
* The child's legal guardian signed the informed consent to participate in the study.
* The legal guardian of the child commits to follow the study procedures and cooperate with the entire study process

Exclusion Criteria:

* Probiotics or antibiotics within 1 month
* Associated with clinically significant abnormalities in liver and kidney function, nervous system, respiratory system, and coagulation function as determined by the investigator
* Unstable vital signs;
* Have other underlying medical conditions
* Individuals deemed unsuitable for this clinical trial.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: heathy children aged 1-3 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiome analysis by high-throughput metagenomic | 0-7 days after enrolled
  The fecal samples from all participants will be collected and subjected to high-throughput metagenomic sequencing in order to elucidate the characteristics and composition of the intestinal microbiome in children residing at different altitudes

SECONDARY OUTCOMES:
Intestinal microbiome metabolites analysis | 0-7 days after enrolled
  This will be detected and analyzed by liquid chromatography-mass spectrometry (LC-MS) non-targeted metabolomics to analyze the metabolites of the intestinal microbiome and compare the differences in these metabolites among children at different altitudes.

OTHER OUTCOMES:
The percentile number of height of children at different altitudes | 0-7 days after enrolled
  Compare the Percentile number of height of children at different altitudes
The percentile number of weight of children at different altitudes | 0-7 days after enrolled
  Compare the Percentile number of weight of children at different altitudes
The percentile number of head circumference of children at different altitudes | 0-7 days after enrolled
  Compare the Percentile number of head circumference of children at different altitudes

CONTACTS AND LOCATIONS:
Overall Officials: Chundi Xu, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China